CLINICAL TRIAL: NCT06434532
Title: An Exploratory Study on the v-Care Interprofessional Online Game for Healthcare Students
Brief Title: Exploring the Effectiveness of an Interprofessional Game-based Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSEARS20230729001
Record Dates: First submitted 2024-01-24; First posted 2024-05-30 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-01

CONDITIONS: Educational Problems
Keywords: Interprofession; online game; nursing; multidisciplinary education

STUDY DESIGN:
Intervention Model Description: waitlist control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- v-Care online game (Experimental): the v-Care online game consist of a clinical scenario. Participants are requested to join the online game in small groups, consisting of nursing and radiography students, to discuss the patient's condition presented in the scenario. They will also be required to watch relevant mini-videos that cover the knowledge check points within the game.
  As part of the activity, participants will be expected to submit a mini interprofessional project that explains their respective roles and responsibilities in managing the patient's condition.
  To enhance engagement and motivation, an online game reward system has been implemented. This system includes the opportunity to earn badges upon completing the knowledge check points or participating in learning activities such as watching tutorials or engaging in interprofessional discussions. These discussions will be recorded and summarized to highlight the key points of their conversation.
  Interventions: Other: v-Care Online Game
- Case-based online discussion (Active Comparator): Participants are requested to engage in case-based discussions within small groups, comprising nursing and radiography students. As part of this activity, students are required to complete a conventional assignment using a worksheet, which will allow them to elaborate on their individual roles and responsibilities in managing the patient's condition.
  In addition, students are encouraged to utilize traditional learning and teaching methods by reading and exploring relevant materials pertaining to the patient's condition.
  Interventions: Other: Case-based online discussion

INTERVENTIONS:
Other: v-Care Online Game — A regular 2 hours traditional learning mode session - case study session and 2-hour online game session with peer-led discussion and interprofessional project submission. This spreads in 3 weeks interval
  Arms: v-Care online game
Other: Case-based online discussion — A 2-hour traditional learning mode session with online peer-led discussion and submission of an interprofessional worksheet as an assignment
  Arms: Case-based online discussion

SUMMARY:
The goal of this waitlist control study is to evaluate the benefits of online game pedagogy to evaluate the readiness of health care students for interprofessional learning in nursing students.

Interprofessional (IP) collaboration is a core competence of health care education to enable effective teamwork and improve health outcomes. Taking into account the characteristics of our students and the pragmatic issues, v-Care (Virtual Care) is a novel strategy to deliver Interprofessional Education using gamification. Colleagues from nursing (SN), rehabilitation sciences (RS) and health technology and informatics (HTI) will collaborate in the design of v-Care, and implement and evaluate it effectiveness in nursing, physiotherapy and radiography related subjects.

To evaluate the effectiveness of interprofessional learning of the health faculty students using a multi-player point-and-click on line motivational game.

Theoretical Framework The v-Care design is based on the Self-Determination Theory (SDT) and Motivational Gamification.

Outcomes:

The primary outcome is to improve the readiness for interprofessional learning. A peer learning community will be established to improve the motivation to learn based on SDT: (1) autonomy, (2) competence and (3) relatedness.

DETAILED DESCRIPTION:
BACKGROUND lnterprofessional education is a core competence of health care education to enable effective collaboration and improve health outcomes [1] (lnterprofessional Education Collaborative Expert Panel, 2011). Numerous initiatives were implemented, including the Freshman Seminar for Broad Disciplines in Health Science (FS) in the undergraduate curriculum. IPE was explicitly listed in the FS intended learning outcomes to (1) understand the professional identity of the learners' own discipline and the other professional's roles on the health care team; and (2) Identify innovative strategies in managing selected major health issues implement using an interprofessional (IP) collaborations approach; and (3) reflect on the experience on interprofessional learning and its implications on lifelong learning and career development. Starting from 2002/23 academic year, this subject was replaced by artificial intelligence and data analytics (AIDA). Since IP is an integral part of the curriculum, implementing IPE under other teaching modes (such as gamification, peer-learning or learner-directed) must be reconsidered.

Motivational gamification is a strategy rooted in the Self-Determination Theory (SDT), gamification and micro-learning are the merits much preferred by the millennials in learning. This strategy leverages on the millennial characteristics that technology has been embedded to their daily life, they enjoy fun and games and are motivated by immediate positive rewards, such as points and badges. Furthermore, they have relatively shorter attention span and enjoy simulation in virtual environments with high quality visuals and graphics. Game features such as click-to-reveal, drag-and-drop, pop quizzes tend to engage the millennial learners. As such, the proposed project is feasible to improve the learning experience and possibly learning outcomes.

AIM To evaluate the effectiveness and impact of interprofessional learning of health faculty students using a multi-player point-and-click on line motivational game. A pretest-posttest non-equivalent waitlist control group design was employed.

METHOD Convenience sampling was adopted to recruit subjects. Inclusion criteria - Participants were recruited from the students who had enrolled in the nursing, physiotherapy and radiography subjects. Students retaking the subject will be excluded from the study.

They were assigned into two study groups according to the tutorial teaching schedule: the control and the experimental groups. The Control group attended the usual teaching activities: paper case study, whereas the intervention group participated in the vCare eGame (intervention). Surveys will be implemented before any learning activities, and at the same time for both groups after the intervention group completed the vCare eGame.

OUTCOME MEASURES Primary outcome will be measured by the Readiness for Interprofessional Learning Scale (19-items).

Secondary outcome on students' autonomy will be measured by a 24-items Perceived Peer Autonomy Support Scale and the 18-item Intrinsic Motivation Inventory.

ELIGIBILITY:
Inclusion Criteria:

* All students learning colorectal cancer and or frailty when taking the specified subject in the Bachelor Nursing Programme and,
* all students taking Bachelor of Science (Honours) Scheme in Medical Laboratory Science and Radiography in Radiography will be recruited

Exclusion Criteria:

* Students retaking these specified subjects will be excluded.
* Students learning other disorders but not colorectal cancer or frailty are not eligible

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Readiness of Health Care Students for Interprofessional Learning (RIPLS) | This will be administered immediately before the start of the learning activity and immediately after the activity is completed
  A 5-point Likert scale questionnaire will be used. There are four subscales that included teamwork and collaboration, negative professional identity, positive professional identity, and roles and responsibility. The higher scores mean a better outcome.

SECONDARY OUTCOMES:
Intrinsic Motivation Inventory | This will be administered immediately before the start of the learning activity and immediately after the activity is completed
  This is a 9-items instrument with 3 subscales: interest/enjoyment, perceived competence, and pressure/tension; on a 7-point Likert Scale - Not at all true, somewhat true to very true.
  The higher scores mean a better outcome
Perceived Autonomy Scale | This will be administered immediately before the start of the learning activity and immediately after the activity is completed
  One 6-items scale will be used to assess the perceive autonomy after the students have completed the learning activity. This is rated on a 7-point Likert Scale - from 1 strongly disagree to 7 strongly agree.
  The higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Kitty Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - School of Nursing, Hung Hom, Hong Kong Island
  - The Hong Kong Polytechnic University, Hung Hom, Hong Kong Island

IPD SHARING:
Plan to Share IPD: Yes
Once the project is completed, and paper published, we are happy to share the IPD.
Supporting Information: Study Protocol, CSR
Time Frame: When the project is completed and publication available
Access Criteria: access by sending email to the corresponding author